CLINICAL TRIAL: NCT00638157
Title: A Phase 4 Multicenter, Randomized, Double Blind Study to Describe the Efficacy and Safety of Cubicin® (Daptomycin for Injection) With and Without Initial Gentamicin Combination Therapy in the Treatment of S. Aureus Infective Endocarditis
Brief Title: Phase 4 Efficacy and Safety Study of Cubicin® With and Without Combination Therapy in S. Aureus Infective Endocarditis (SAIE)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: commitment completed
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3009-010; DAP-4IE-06-03 (Other: Cubist Study Number)
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Infective Endocarditis
Keywords: Gram-positive bacterial infections; Staph Aureus; endocarditis; bacteremia; methicillin-resistant Staphylococcus aureus (MRSA)
MeSH Terms: conditions — Endocarditis; Gram-Positive Bacterial Infections; Staphylococcal Infections; Bacteremia | interventions — Daptomycin; Injections; Gentamicins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daptomycin Alone (Active Comparator): daptomycin 6 mg/kg q24h for treatment of right-sided infective endocarditis
  Interventions: Drug: daptomycin
- Daptomycin plus gentamicin (Experimental): daptomycin 6 mg/kg q24h with concomitant initial gentamicin dosed for the first 2 days of therapy for the treatment of right-sided infective endocarditis
  Interventions: Drug: daptomycin and gentamicin

INTERVENTIONS:
Drug: daptomycin — Intravenous (i.v.) 6 mg/kg q24h
  Other Names: Cubicin; daptomycin for injection
  Arms: Daptomycin Alone
Drug: daptomycin and gentamicin — i.v. daptomycin 6 mg/kg q24h plus initial i.v. gentamicin
  Other Names: Cubicin; daptomycin for injection; gentamicin
  Arms: Daptomycin plus gentamicin

SUMMARY:
multicenter, randomized, double blind study to describe the safety and efficacy of daptomycin (6 mg/kg q24h) with and without concomitant initial gentamicin combination therapy in the treatment of SAIE

DETAILED DESCRIPTION:
Patients will be randomized to either of the following two treatment arms:

* Arm 1: daptomycin
* Arm 2: daptomycin with initial i.v. gentamicin

Patients who meet all the inclusion criteria and exhibit none of the exclusion criteria may be enrolled. Intravenous drug user (IVDU) patients may be randomized and study drug begun on the basis of two separate peripheral blood cultures positive for S. aureus obtained within 96 hours prior to the first dose of study drug.

The recommended minimum duration of treatment for daptomycin will be 28 days. The duration of treatment for gentamicin will be 3 days.

During study treatment, regular assessments (including weekly safety laboratory testing including CPK) will be performed. An End-of-Therapy (EOT) evaluation will be performed on the day of or 1-2 days after completion of daptomycin study drug or upon early termination (ET). All patients will have a post-therapy visit for Test of Cure (TOC)/Safety performed 21-28 days following the last dose of daptomycin study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained;
2. Male or female ≥18 years of age;
3. IVDU (as confirmed by history of drug abuse within the past 3 months or recent needle track marks);
4. Definite or possible IE according to the modified Duke Criteria (see Appendix A); [17 ];
5. Two blood cultures positive for S. aureus obtained within 96 hours prior to first dose of study medication acquired by fresh venipuncture using aseptic technique and analyzed at the local laboratory (see Appendix B).

Exclusion Criteria:

1. Intravascular foreign material in place at the time that the positive blood culture was drawn (e.g., intracardiac pacemaker wires, percutaneous or implanted venous catheters, vascular grafts), (exception: vascular stents that have been in place for >6 months or permanent pacemaker wires attached via epicardial leads are allowed);
2. High likelihood of LIE as indicated by:

   1. Prior diagnosis of predisposing left-sided valvular pathology (e.g., rheumatic heart disease, bicuspid aortic valve); or
   2. Findings on screening examination of left-sided valvular pathology (e.g., diastolic murmur of aortic insufficiency); or
   3. Findings on screening examination of major systemic emboli to visceral organs (e.g. cerebral or splenic infarct). Patients may be included if their only findings are consistent with microvascular phenomena due to immune complexes (e.g., splinter hemorrhages, conjunctival petechiae, Roth's spots, Osler's nodes, Janeway's lesions, microhematuria).

   Note: Any patient enrolled in the study that is subsequently found to have LIE may be continued in the trial if determined to be clinically improving by the Investigator.
3. Prosthetic heart valve;
4. Baseline Creatinine clearance of <30 mL/min (as calculated by the Cockcroft-Gault equation using actual body weight);
5. Baseline CPK value 5 X upper limit of normal (ULN) in conjunction with symptoms of myalgia or baseline CPK value 10 X ULN without symptoms;
6. Alanine aminotransferase (ALT) >5 X ULN;
7. Aspartate aminotransferase (AST) >5 X ULN;
8. Moribund clinical condition (i.e. high likelihood of death within 3 days after randomization);
9. Shock or hypotension (supine systolic blood pressure <80 mm Hg) or oliguria (urine output <20 mL/h) unresponsive to fluids or pressors within 4 hours;
10. Known pneumonia or osteomyelitis;
11. Polymicrobial infection or bacteremia due to a pathogen other than S. aureus;
12. Neutropenia (absolute neutrophil count < 0.5 X 103/μL) and/or lymphopenia (CD4 lymphocytes <0.2X 103/μL);
13. Anticipated to require non-study antibiotics that may be potentially effective against S. aureus;
14. Prior gentamicin therapy > 1 day;
15. Documented history of significant allergy or intolerance to any of the study medications;
16. Unlikely to comply with study procedures;
17. Pregnant or nursing. All females with childbearing potential will have a pregnancy test performed at the local laboratory.
18. Female of childbearing potential and not willing to practice barrier methods of birth control (e.g., condoms or diaphragms together with spermicidal foam or gel) during treatment and for at least 28 days after treatment with study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02-13 (Actual); Primary Completion 2011-11-09 (Actual); Study Completion 2011-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Bokesch, M.D., Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (4):
- United States (4):
  - Denver Health Medical Center, Denver, Colorado
  - Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Temple University School of Medicine, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Daptomycin: Intravenous daptomycin 6mg/kg every 24 hours for a recommended minimum duration of 28 days plus a
- Daptomycin Plus Gentamicin: Intravenous daptomycin 6mg/kg every 24 hours for a recommended minimum duration of 28 days plus intravenous gentamicin 1mg/kg every 8 hours for the first 3 days of daptomycin therapy.
Period: Overall Study
Arm/Group | Daptomycin | Daptomycin Plus Gentamicin
Started | 12 | 12
Treated | 10 | 12
Completed | 5 (4 subjects completed study drug in this arm) | 8 (4 subjects completed study drug in this arm)
Not Completed | 7 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Clinical (symptomatic) failure | 1 | 1
Not completed — Microbiological failure | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Other | 1 | 2
Not completed — Randomized, not treated | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population used. Includes all randomized subjects.
Groups:
- Daptomycin: Intravenous daptomycin 6mg/kg every 24 hours for a recommended minimum duration of 28 days plus a "dummy" infusion of 0.9% normal saline every 8 hours for the first 3 days of daptomycin therapy.
- Total: Total of all reporting groups
Arm/Group | Daptomycin | Daptomycin Plus Gentamicin | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (10.93) | 45.3 (9.90) | 42.1 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Summary of Clinically Significant Increases in Serum Creatinine by Visit
Description: The End of Treatment (EOT)/Early Termination (ET) visit occurred on the day that therapy was stopped or up to 2 days after the last dose of daptomycin. The Test of Cure (TOC)/Safety visit occurred 21 to 28 days after the last dose of daptomycin therapy. The overall median duration of treatment was 13.0 days in both the daptomycin group and the combination therapy group. The definition of elevated serum creatinine at baseline is >3.0 mg/dL, and not elevated is ≤3.0 mg/dL. Clinically significant increases in serum creatinine is defined as an increase ≥0.5 mg/dL for patients with a baseline value ≤3.0 mg/dL or ≥1.0 mg/dL for patients with a baseline value >3.0 mg/dL.
Time Frame: Baseline, EOT Visit, TOC
Population: Safety Population includes all patients who received any dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Daptomycin | Daptomycin Plus Gentamicin
Number analyzed (Participants) | 10 | 12
Participants
  Baseline - Any Elevation | 0 | 0
  Baseline - No Elevation | 10 | 12
  End of Therapy - Any Elevation | 0 | 2
  End of Therapy - No Elevation | 10 | 10
  Test of Cure - Any Elevation (n=8,9) | 0 | 2
  Test of Cure - No Elevation (n=8,9) | 8 | 7

2. Secondary Outcome: Summary of the Investigator's Assessment of Clinical Response at the TOC Visit
Description: TOC/Safety visit occurred 21 to 28 days after the last dose of daptomycin therapy. Clinical response was assessed by the investigator as cure, improvement, failure, and unable to evaluate. Microbiological response, which was determined by the sponsor based on review of baseline and post-baseline culture results, included success, failure, and nonevaluable. TC=Treatment Cure; TF=Treatment Failure; TI=Treatment Improved.
Time Frame: TOC Visit
Population: Modified Intent-to-Treat (mITT) population includes all ITT patients who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Daptomycin | Daptomycin Plus Gentamicin
Number analyzed (Participants) | 9 | 11
Participants
  TC (clinical cure, microbiological success) | 4 | 5
  TC (clinical cure, microbiological nonevaluable) | 0 | 0
  TF (clinical failure, microbiological success) | 1 | 1
  TF (clinical cure, microbiological failure) | 0 | 0
  TF (clinical failure, microbiological failure) | 2 | 0
  TF (clinical improved, microbiological failure) | 0 | 0
  TF (clinical failure, microbiological nonevaluable | 0 | 2
  TI (clinical improved, microbiological success) | 0 | 1
  TI (clin improved, microbiological nonevaluable) | 0 | 0
  Non-evaluable | 2 | 2

ADVERSE EVENTS:
Arm/Group | Daptomycin | Daptomycin Plus Gentamicin
Serious Adverse Events (participants affected / at risk) | 2/10 | 5/12
Other Adverse Events (participants affected / at risk) | 8/10 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daptomycin (N=10) | Daptomycin Plus Gentamicin (N=12)
Tachycardia (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daptomycin (N=10) | Daptomycin Plus Gentamicin (N=12)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Abnormal sensation in eye (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 2
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Catheter related complication (General disorders) | 3 | 1
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 4 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
As the study was terminated prematurely, conclusions that can be drawn from the efficacy results are limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication is initiated by Cubist. If First Publication not published within 1 year of Study conclusion or termination, Investigator has right to publish and disclose the Data. Prior to any submission for publication, presentation, or communication of results or information arising from the Study, Investigator shall provide Cubist at least 90 days for review and comment upon the manuscript or other material for such publication or presentation.